CLINICAL TRIAL: NCT03090412
Title: A Randomized Multicenter Phase II Study Using (2-1[Heyloxyethyl]-2-Devinylpyropheophorbide-a) (HPPH) With PDT Versus Standard of Care Surgery for Patients With T1/T2 N0 Squamous Cell Carcinoma of the Oral Cavity
Brief Title: Photodynamic Therapy With HPPH Compared to Standard of Care Surgery in Treating Patients With Oral Cavity Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 33616; NCI-2017-00441 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 33616 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2017-03-20; First posted 2017-03-24 (Actual); Results first posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Stage I Oral Cavity Squamous Cell Carcinoma; Stage II Oral Cavity Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — 2-(1-hexyloxyethyl)-2-devinyl pyropheophorbide-a; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Phototherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (surgery) (Experimental): Patients undergo standard of care surgery on day 1.
  Interventions: Other: Quality-of-Life Assessment; Procedure: Therapeutic Conventional Surgery
- Arm II (HPPH, PDT) (Experimental): Patients receive HPPH IV over 1 hour on day 0 and undergo PDT on day 1.
  Interventions: Drug: HPPH; Other: Laboratory Biomarker Analysis; Drug: Photodynamic Therapy; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: HPPH — Given IV
  Other Names: Photochlor
  Arms: Arm II (HPPH, PDT)
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Arm II (HPPH, PDT)
Drug: Photodynamic Therapy — Undergo PDT
  Other Names: PDT; Photoradiation Therapy
  Arms: Arm II (HPPH, PDT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Procedure: Therapeutic Conventional Surgery — Undergo standard of care surgery
  Arms: Arm I (surgery)

SUMMARY:
This randomized phase II clinical trial studies how well photodynamic therapy with HPPH works compared to standard of care surgery in treating patients with oral cavity cancer. Photodynamic therapy can destroy or control disease by using a combination of drug, such as HPPH, and light and may be as effective as surgery in treating patients with oral cavity cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the non-inferiority of photodynamic therapy (PDT) to standard of care surgery by comparing the rate of tumor response after PDT to those observed after surgery, at 24 months post treatment.

SECONDARY OBJECTIVES:

I. To determine quality of life (QoL) at 6, 12, 18 and 24 months post PDT or surgery.

II. To assess the toxicity using the Cancer Therapy Evaluation Program (CTEP) National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE Version 4.0).

TERTIARY OBJECTIVES:

I. Immune markers (T cells). II. To investigate the correlation of the diffuse reflectance optical spectroscopy with tumor response to PDT.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo standard of care surgery on day 1.

ARM II: Patients receive HPPH intravenously (IV) over 1 hour on day 0 and undergo PDT on day 1.

After completion of study treatment, patients are followed up every 3-4 months in year 1 and every 3-6 months in year 2.

ELIGIBILITY:
Inclusion Criteria:

* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Participants with previously untreated T1/T2 N0 squamous cell carcinoma of the oral cavity with or without extension to the oropharynx
* Histologically confirmed squamous cell carcinoma of the target tumor(s)
* Tumor thickness is 4 mm or less (measured clinically and/or by computed tomography [CT] or magnetic resonance imaging [MRI] scan)
* CT or MRI of the neck to confirm staging
* Tumor accessible for unrestricted illumination for photodynamic therapy (PDT) (accessibility as determined by the physician)
* Life expectancy of at least 12 months in the judgment of the physician
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Participant or legal representative must understand the investigational nature of this study and sign an Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Those who have had chemotherapy or radiotherapy or targeted agents within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Those with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Those with porphyria or with known hypersensitivity to porphyrins or porphyrin-like compounds
* White blood cells (WBC) < 4,000
* Total serum bilirubin > 2 mg/dL
* Serum creatinine > 2 mg/dL
* Alkaline phosphatase (hepatic) or serum glutamic-oxaloacetic transaminase (SGOT) > 3 times the upper normal limit
* Diagnostic biopsy reveals perineural invasion (PNI) and/or lymphovascular invasion (LVI)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Nodal disease as detected by clinical exam or CT
* Pregnant or nursing females
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Received an investigational agent within 30 days prior to enrollment
* Trismus or compromised airway
* Previous treatment in the target tumor area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Chan, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rocherster, Rochester, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Surgery) | Arm II (HPPH, PDT)
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Surgery) | Arm II (HPPH, PDT) | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 86 [86 to 86] | 55 [55 to 55] | 71 [55 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Tumor Response as Evaluated by Response Evaluation Criteria in Solid Tumors Version 1.1
Description: Objective tumor response will be tabulated overall.
Time Frame: At 24 months
Population: Due to PI departure and early termination with few patients, only the counts of events have been calculated and no testing was done
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Surgery) | Arm II (HPPH, PDT)
Number analyzed (Participants) | 1 | 1
Participants
  No evidence of disease | 1 | 0
  Other | 0 | 1

2. Secondary Outcome: Change in Quality of Life as Measured by the University of Washington Quality of Life Questionnaire Version 4
Description: In the analysis of QoL simple data analyses will initially take place including individual participant-level profile plots and overall mean plots used to examining the mean structure. Formal statistical examination of longitudinal patterns will be done through the use of a mixed model. Once the model is fit, specific linear contrasts based on the estimated model parameters will be constructed and used to test hypotheses concerning between time points and between group comparisons
Time Frame: Baseline up to 24 months
Population: Due to PI departure with few patients, only the counts of events have been calculated and no testing was done..
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Surgery) | Arm II (HPPH, PDT)
Number analyzed (Participants) | 1 | 1
Participants
  Outstanding Overall QoL | 1 | 0
  Very good to Outstanding Overall QoL | 0 | 1

3. Secondary Outcome: Adverse Events as Graded by CTCAE Version 4.0 Are Reported
Description: The frequency of toxicities will be tabulated by grade.
Time Frame: Up to 30 days after administration of HPPH
Population: Due to PI departure with few patients, only the counts of events have been calculated and no tabulation was done..
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Surgery) | Arm II (HPPH, PDT)
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: From administration of study drug or surgery until 30 days after receiving study drug or surgery
Arm/Group | Arm I (Surgery) | Arm II (HPPH, PDT)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Surgery) (N=1) | Arm II (HPPH, PDT) (N=1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Surgery) (N=1) | Arm II (HPPH, PDT) (N=1)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue exfoliation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT03090412/Prot_SAP_000.pdf